CLINICAL TRIAL: NCT02420470
Title: The Early Warning System for the Central Nervous System Micro-structure Alterations During Early Diabetes Based on the Multi-mode MRIs
Brief Title: The Early Warning System for the Diabetic Encephalopathy
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDLL-2014086
Record Dates: First submitted 2015-04-02; First posted 2015-04-17 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus Type 2; Mild Cognitive Impairment; Metabolic Syndrome X
Keywords: diabetes; neural and vessel alteration; prodromal stage
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Metabolic Syndrome; Diabetes Mellitus; Prodromal Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy control group: fasting plasma glucose(FPG)<6.11mmol/L，and 2-h plasma glucose(2hPG)<7.77mmol/L；
- prodromal diabetes group: IFG：fasting plasma glucose(FPG) ≥5.6mmol/L (100mg/dl)，and<7.0mmol/L (126mg/dl)，oral glucose tolerance test(OGTT) 2-h plasma glucose(2hPG) <7.8 mmol/L ；IGT：oral glucose tolerance test(OGTT) 2-h plasma glucose(2hPG) ≥7.8mmol/L (140mg/dl)，and<11.1mmol/L (200mg/dl)，fasting plasma glucose(FPG)< 5.6mmol/L
- diabetes group: fasting plasma glucose(FPG)>7.0mmol/L, or 2-h plasma glucose(2hPG)>11.1mmol/L

SUMMARY:
Diabetes( mainly type II diabetes )lead to the central nervous system (CNS) function impairment, especially the mild cognitive impairment that increased the risk of progression to dementia.The primary objectives are defined according to a hierarchical design: i) to tailor and apply multi-parametric, functional MRI techniques to identify cerebral abnormalities (cerebral biomarkers) in type 2 diabetes mellitus and prodromal diabetes mellitus ; ii) to assess whether these cerebral biomarkers are associated with cognitive decrements;iii) to follow up with the putative prediabetic condition patients to verify whether they can transform into diabetes.

DETAILED DESCRIPTION:
Diabetes ( mainly type II diabetes ) lead to the central nervous system (CNS) function impairment, especially the mild cognitive impairment (MCI) that increased the risk of progression to dementia. It was regarded that neurodegeneration contributes to the diabetic MCI, however, recent research suggested that CNS microvascular alterations are the mechanism for early diabetic MCI. But there still lacks an early warning system for the CNS micro-structure alterations during early diabetes. Latest neuroimaging techniques enable the measurement of brain blood flow, local neural activity，and the nuclei deposition of iron to reflect CNS micro-structure alterations. But these techniques are complicated and can not fully reflect the alterations with one single technique.We previous observed that 44.4% of diabetic patients demonstrate MCI and established the comprehensive protocols of measuring brain blood flow, local neural activity and the nuclei deposition of iron simultaneously based on the multimodal MRI technique so as to reflect the microstructure alterations reliably and validly. Therefore, we intend to integrate psychological measurement and clinical biochemical examination, and to establish the early warning system for the central nervous system micro-structure alterations during early diabetes based on the multi-modal MRI technique. The reliability and validity of this system will be tested in the diabetic rat model. The early warning system will likely assist in screening patients with diabetic microstructure alterations, to perform early intervention so as to prevent or delay the progression from diabetic MCI to dementia.

ELIGIBILITY:
Inclusion Criteria:

* without dementia
* Inform Consent Form
* Education time more than 6 years
* blood glucose matches the group standard

Exclusion Criteria:

* Pregnant woman
* suffer from serious brain disease
* Magnetic resonance contraindications
* lack of compliance
* image quality is too poor to deal with

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: prodromal diabetes and early diabetes
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional and structural connectivity relationships of multiple brain regions and biomarkers of brain alterations, and the changes in relationships and biomarkers at 2.5 years. | subjects will be assessed six times (once half a year, up to 2.5 years )
  Differences in macro-structural and micro-structural between patients,prodromal group and healthy controls will be evaluated. These MRI measures include volumetric characteristics (e.g. hyper-intensities, white matter lesions, atrophy, cerebral microbleeds), quantitative measures (e.g. T2 relaxation times, mean diffusivity, fractional anisotropy, mean kurtosis), functional characteristics (e.g. activated regions, cerebral blood flow), network properties (e.g. functional and structural connectivity, graph-theoretical measures).

SECONDARY OUTCOMES:
evaluation of obesity and the changes in the state of obesity at 2.5 years | subjects will be assessed six times (once half a year, up to 2.5 years)
  Simple evaluation of obesity will include: Body mass index will be calculated as the weight (kg) divided by the square of the height (m). Waist circumference (WC) will be taken as the minimum circumference between the umbilicus and xiphoid process and measured to the nearest 0.5 cm.
metabolic characteristics and their changes at 2.5 years | subjects will be assessed six times (once half a year, up to 2.5 years)
  Simple metabolic characteristics will include: oral glucose tolerance test, C peptide releasing test and insulin releasing test will be assessed;homeostasis model assessment of insulin resistance，insulin secretion of homeostasis model assessment and homeostasis model assessment-β will be calculated. what's more, cardiovascular risk factors(e.g. albumin, creatinin, total cholesterol, LDL- and HDL-cholesterol, triglycerides, HbA1c) will be assessed.
Mental health and the changes in the scores of the scales at 2.5 years | subjects will be assessed six times (once half a year, up to 2.5 years)
  To evaluate the mental health, a series of psychiatric evaluation scale(e.g. mini-mental state examination, Montreal Cognitive Assessment，Hamilton anxiety scale, self-rating depression scale, frontal assessment battery) will be assessed.
Lifestyle and its changes at 2.5 years | subjects will be assessed six times (once half a year, up to 2.5 years)
  Lifestyle specifics, including alcohol consumption, smoking behavior and mobility and exercise habit will be obtained. At the same time, quality of life will be obtained through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Guangbin Cui, professor, Study Chair — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Hu B, Yu Y, Yu XW, Ni MH, Cui YY, Cao XY, Yang AL, Jin YX, Liang SR, Li SN, Dai P, Wu K, Yan LF, Gao B, Cui GB. Sequence of episodic memory-related behavioral and brain-imaging abnormalities in type 2 diabetes. Nutr Diabetes. 2025 Feb 1;15(1):1. doi: 10.1038/s41387-025-00359-w. PMID 39893169
- [Derived] Hu B, Yan LF, Sun Q, Yu Y, Zhang J, Dai YJ, Yang Y, Hu YC, Nan HY, Zhang X, Heng CN, Hou JF, Liu QQ, Shao CH, Li F, Zhou KX, Guo H, Cui GB, Wang W. Disturbed neurovascular coupling in type 2 diabetes mellitus patients: Evidence from a comprehensive fMRI analysis. Neuroimage Clin. 2019;22:101802. doi: 10.1016/j.nicl.2019.101802. Epub 2019 Mar 27. PMID 30991623
- [Derived] Sun Q, Chen GQ, Wang XB, Yu Y, Hu YC, Yan LF, Zhang X, Yang Y, Zhang J, Liu B, Wang CC, Ma Y, Wang W, Han Y, Cui GB. Alterations of White Matter Integrity and Hippocampal Functional Connectivity in Type 2 Diabetes Without Mild Cognitive Impairment. Front Neuroanat. 2018 Mar 20;12:21. doi: 10.3389/fnana.2018.00021. eCollection 2018. PMID 29615873
- [Derived] Yu Y, Sun Q, Yan LF, Hu YC, Nan HY, Yang Y, Liu ZC, Wang W, Cui GB. Multimodal MRI for early diabetic mild cognitive impairment: study protocol of a prospective diagnostic trial. BMC Med Imaging. 2016 Aug 24;16(1):50. doi: 10.1186/s12880-016-0152-x. PMID 27552827